CLINICAL TRIAL: NCT03365440
Title: Esophageal 3D Mapping System for Cardiac Arrhythmias: Pilot Study to Establish Basis for Improved Arrhythmia Diagnostics Using the esoECG-3D Catheter
Brief Title: Esophageal 3D Mapping System for Cardiac Arrhythmias
Acronym: esoECG-3D
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: CR23I2_166030
Record Dates: First submitted 2017-10-26; First posted 2017-12-07 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Arrhythmia; Atrial Fibrillation; Atrial Flutter; Atrial Tachycardia; Supraventricular Tachycardia; Ventricular Ectopic Beat(S); Cardiac Arrythmias
Keywords: ECG; cardiac arrhythmia; heart rhythm; esophageal ECG; non-invasive mapping; supraventricular tachycardia; atrial fibrillation; atrial flutter; extrasystole
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation; Atrial Flutter; Tachycardia, Supraventricular; Ventricular Premature Complexes; Cardiac Complexes, Premature

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- EP study with transseptal passage: * 15-30 minute esophageal ECG (using esoECG-3D catheter) & respiration recording during elective EP study and/or ablation procedure
  * Focal pacing maneuvers
  Interventions: Device: esoECG-3D catheter
- EP study without transseptal passage: - 15-30 minute esophageal ECG (using esoECG-3D catheter) & respiration recording during elective EP study and/or ablation procedure
  Interventions: Device: esoECG-3D catheter
- Healthy participants: - 60 minute esophageal ECG (using esoECG-3D catheter) & respiration recording
  Interventions: Device: esoECG-3D catheter

INTERVENTIONS:
Device: esoECG-3D catheter — Recording of esophageal ECGs with the investigational medical device (IMD). Recording of respiration with a commercial breathing sensor.

SUMMARY:
The aim of the study is to develop and validate a novel esophageal mapping system to improve the diagnostics of cardiac arrhythmias. Using a newly designed esophageal ECG catheter, esophageal ECGs (eECGs) will be recorded in 40 patients during an electrophysiological (EP) study and/or ablation procedure and in 12 healthy volunteers. In parallel acquired intracardiac electrograms will serve as reference for the developed mapping systems accuracy. Additionally, the esophageal mapping system will be compared to that of the standard 12-lead surface ECG in regard to its diagnostic performance.

DETAILED DESCRIPTION:
Background

Cardiac arrhythmias are common and may have devastating consequences for affected patients. To prevent f.e. strokes due to atrial fibrillation, heart failures as a consequence of long-standing tachyarrhythmias or death due to ventricular fibrillation, accurate and timely diagnoses are essential. The standard diagnostic tool for heart rhythm disorders in everyday clinical life is the 12-channel surface electrocardiogram (ECG). However, despite its strengths, the surface ECG suffers from several limitations. Especially on the supraventricular level, the low atrial signal amplitude renders it prone to errors and causes surface ECGs to quickly reach the limits of their diagnostic capacities.

This limitation could be overcome by recordings through the esophagus. Owing the close anatomical relationship, esophageal ECGs have an excellent atrial signal quality. To fully exploit their potential, a novel esophageal ECG catheter (esoECG catheter) with 3-dimensional electrode arrangement was developed. The aim of this study is to use the esoECG-3D catheter to develop and validate a non-invasive esophageal mapping system in order to improve the diagnostics of cardiac arrhythmias and consequently the therapy of patients suffering from these disorders.

Objectives

Primary objective (A1): Development of an esophageal non-invasive mapping system which shall be able to depict

* A1.1: the source of focal triggers
* A1.2: the sequence of cardiac depolarization

with high spatial and temporal resolution.

Secondary objectives (A2):

* A2.1: outperform the diagnostic accuracy of 12-lead ECGs in bedside arrhythmia diagnostics
* A2.2: estimate the speed of myocardial depolarization on the left atrial wall from esophageal ECG tracings
* A2.3: extract respiration signals from esophageal ECG tracings
* A2.4: determine the wearing comfort of the device
* A2.5: determine the operability of the device

Safety objective (A3): Determination of safety of the esoECG-3D catheter for esophageal ECG recordings with respect to:

* A3.1: device related adverse events
* A3.2: device related serious adverse events
* A3.3: device failures, including insertion failure

Methods

Esophageal ECGs will be acquired from a total of 52 participants using the esophageal esoECG-3D catheter. 40 of these will be recorded during an electrophysiological study and/or ablation procedure to obtain a reference (intracardiac measurements) for the evaluation of outcome measures. In a subset of patients, defined pacing maneuvers will be performed; 12-channel ECG and breathing sensor recordings will be obtained from all participants in parallel to eECG measurements. The acquired data will be used for development of algorithms to non-invasively map the hearts depolarization process from recordings in the esophagus. Outcome evaluation will be performed after completion of all measurements and after implementation of the final mapping algorithms.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* Age >18 years
* Group 1: Patients scheduled for an elective electrophysiological study and/or ablation procedure including a transseptal passage
* Group 2: Patients, scheduled for an elective electrophysiological study and/or ablation procedure without transseptal passage
* Group 3: Healthy volunteers, without any known cardiac disease

Exclusion Criteria:

* Contraindications to the class of devices under study, e.g. known hypersensitivity or allergy to class of devices or the investigational device
* Status post atrial fibrillation ablation within the last 4 weeks
* Unstable angina pectoris or acute coronary syndrome
* Hemodynamic instability
* Respiratory instability
* Disease or malformation of the upper airways or esophagus, making naso-esophageal catheter insertion impossible
* Hereditary severe bleeding diathesis
* Status post surgical intervention of the esophagus or stomach within the last 4 weeks
* Known cancer of the esophagus or stomach
* Pregnancy
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of (40) adult patients that are scheduled for an elective electrophysiological study and/or ablation procedure at the study location and of (12) healthy volunteers without any known heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of focal trigger localization by esophageal mapping system | within 1 year after study completion
  Reference: intracardiac recordings
Accuracy of cardiac activation sequence estimation by esophageal mapping system | within 1 year after study completion
  Reference: intracardiac recordings

SECONDARY OUTCOMES:
Diagnostic performance of esophageal mapping system compared to standard 12-channel ECG | within 1 year after study completion
  Reference: intracardiac recordings
Accuracy of depolarization propagation speed estimation from eECGs (acquired with IMD) | within 1 year after study completion
  Reference: intracardiac recordings
Accuracy of respiration estimation from eECGs (acquired with IMD) | within 1 year after study completion
  Reference: breathing sensor recordings
Incidence of Adverse Events [Safety and Tolerability] | up to 12 hours after study completion
  Incidence of Treatment-Emergent Adverse Events to determine safety and tolerability of IMD

CONTACTS AND LOCATIONS:
Overall Officials: Hildegard Tanner, MD, Principal Investigator — Department of Cardiology, University Hospital Inselspital Bern
Locations (1):
- Department of Cardiology, University Hospital Inselspital Bern, Bern, Canton of Bern, Switzerland